CLINICAL TRIAL: NCT04440501
Title: Virtual Reality to Teach, Improve Outcomes, and Engage (VIRTUE): Virtual Reality to Improve Gluten-Free Diet Knowledge in Pediatric Celiac Disease, A Randomized Clinical Trial
Brief Title: Virtual Reality to Teach, Improve Outcomes, and Engage (VIRTUE): Virtual Reality to Improve Gluten-Free Diet Knowledge in Pediatric Celiac Disease
Acronym: VIRTUE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Nasim Khavari, Clinical Associate Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 56017
Record Dates: First submitted 2020-06-17; First posted 2020-06-19 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Celiac Disease in Children

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard education (Control) (No Intervention): Standard education regarding the gluten free diet by the nutritionist will be provided.
- Virtual Reality Program to teach gluten free diet (Experimental): Virtual Reality Goggles and education regarding the gluten free diet will be provided.
  This group will receive VIRTUE, and watch a VR educational video, and play Chaos Café, which will be administered by a research team member. This group will be prescribed to take home the VIRTUE headset and play modules for 15 minutes per week until the 6-8 month follow up.
  The VIRTUE technology will track frequency of game playing to control for adherence to the prescription.
  Interventions: Device: Virtual Reality Goggles to provide education a regarding the gluten free diet.

INTERVENTIONS:
Device: Virtual Reality Goggles to provide education a regarding the gluten free diet. — To watch and participate in a virtual reality educational experience regarding the gluten free diet.
  Arms: Virtual Reality Program to teach gluten free diet

SUMMARY:
1. Specific Aim (1) is to assess both the immediate and longer term impact of VIRTUE on the patient's GFD knowledge compared to standard of care (SOC) dietary education.
2. Specific Aim (2) is to determine the impact of VIRTUE on patient QoL, symptomatology, and Celiac biomarkers (tissue transglutaminase antibodies, deamidated gliadin peptide IgA, deamidated gliadin peptide IgG, and total serum IgA).

DETAILED DESCRIPTION:
The global burden of Celiac Disease (CD) is estimated to be 1% in Western countries and 0.7-1.4% of the global population.The only treatment for CD is a strict, lifelong Gluten Free Diet (GFD). However, dietary adherence is the main barrier against disease control. Whereas experiential learning, learning through experience, has been associated with greater impact in achieving desired nutritional outcomes in pediatric populations. Replicating the environments in which patients would make food choices in clinic is not feasible.

Previous research, in addition to preliminary results indicate that Virtual reality (VR) may act as an effective precursor to the real world by providing a safe and immersive learning environment. As such, the investigators seek to investigate how VR use to Teach, Improve Outcomes, and Engage (VIRTUE) will affect patient GFD knowledge, QoL, symptoms, and CD biomarkers. The central hypothesis will tested through the following specific aims:

1. Specific Aim (1) is to assess the immediate and long-term impact of VIRTUE on children's GFD knowledge compared to SOC education. The investigators hypothesize that VIRTUE with SOC education, will improve children's GFD knowledge by 10-20%, opposed to SOC alone
2. Specific Aim (2) is to determine the impact of VIRTUE on patient QoL. The investigators hypothesize that VIRTUE with SOC education, will improve children's QoL scores, opposed to SOC alone.
3. Specific Aim (3) is to determine the impact of VIRTUE on decline of CD biomarkers (tissue transglutaminase antibodies and deamidated gliadin peptide IgG). The investigators hypothesize that VIRTUE with SOC education, will reduce levels of CD biomarkers faster, compared to SOC alone.

ELIGIBILITY:
Inclusion Criteria:

* Patients with confirmed diagnosis of CD per American or European Guidelines
* Ages 8-18 years of all genders

Exclusion Criteria:

-Significant Developmental Delays

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-09-28 (Estimated); Primary Completion 2025-03-28 (Estimated); Study Completion 2026-01-28 (Estimated)

PRIMARY OUTCOMES:
Knowledge of the Gluten Free Diet | 9 months
  GFD-KS at the initial and clinic follow up visit

SECONDARY OUTCOMES:
CD Quality of Life | 9 months
  QoL survey
Biomarkers to asses status of GFD | 6-9 months
  Biomarkers maximum value (Ttg IgA and Dgp IgA)

IPD SHARING:
Plan to Share IPD: No